CLINICAL TRIAL: NCT02288481
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study With a Food Effect Cohort to Evaluate the Safety, Tolerability, and Pharmacokinetics of TBA-354 in Healthy Adult Subjects
Brief Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TBA-354 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TBA-354-CL-001
Record Dates: First submitted 2014-11-07; First posted 2014-11-11 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; TBA-354; Pulmonary Tuberculosis; TB
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary | interventions — TBA-354

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- Cohort 1 10 mg TBA-354 (Experimental)
  Interventions: Drug: TBA-354
- Cohort 1 placebo (Placebo Comparator): Placebo Suspension
  Interventions: Other: Placebo
- Cohort 2 25 mg TBA-354 (Experimental)
  Interventions: Drug: TBA-354
- Cohort 2 placebo (Placebo Comparator): Placebo Suspension
  Interventions: Other: Placebo
- Cohort 3 60 mg TBA-354 (Experimental)
  Interventions: Drug: TBA-354
- Cohort 3 placebo (Placebo Comparator): Placebo Suspension
  Interventions: Other: Placebo
- Cohort 4 150 mg TBA-354 (Experimental)
  Interventions: Drug: TBA-354
- Cohort 4 placebo (Placebo Comparator): Placebo Suspension
  Interventions: Other: Placebo
- Cohort 5 400 mg TBA-354 (Experimental)
  Interventions: Drug: TBA-354
- Cohort 5 placebo (Placebo Comparator): Placebo Suspension
  Interventions: Other: Placebo
- Cohort 6 1000 mg TBA-354 (Experimental)
  Interventions: Drug: TBA-354
- Cohort 6 placebo (Placebo Comparator): Placebo Suspension
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TBA-354 — TBA-354 supplied as a 20 mg /mL suspension and matching placebo suspension for oral administration.
  Arms: Cohort 1 10 mg TBA-354; Cohort 2 25 mg TBA-354; Cohort 3 60 mg TBA-354; Cohort 4 150 mg TBA-354; Cohort 5 400 mg TBA-354; Cohort 6 1000 mg TBA-354
Other: Placebo — Placebo Suspension
  Arms: Cohort 1 placebo; Cohort 2 placebo; Cohort 3 placebo; Cohort 4 placebo; Cohort 5 placebo; Cohort 6 placebo

SUMMARY:
The objective of this study is to evaluate the safety and tolerability of single oral doses of TBA-354 when administered to healthy adult subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single ascending dose study conducted at one study center in the United States. Six (6) cohorts of 8 subjects each (6 active and 2 placebo), with one cohort crossing over to assess food effect, are planned for evaluation. Subjects will participate in only one cohort.

Safety will be assessed throughout the study; serial ECGs and serial blood samples will be collected for the safety and PK assessment of TBA-354.

Dose escalation to the next cohort (i.e., dose level) will not take place until the Sponsor, in conjunction with the Principal Investigator, has determined that adequate safety, tolerability and PK from the previous cohort has been demonstrated to permit proceeding to the next cohort. Upon review of cohort data, the Sponsor, in conjunction with the Principal Investigator, may decide to:

1. Escalate dose as planned.
2. Evaluate an intermediate dose level prior to proceeding to the next planned dose level if concerns arise from signs and symptoms that do not warrant ceasing escalation as described above.
3. Repeat a given dose level in a new cohort of subjects.
4. Halt the study.

Blinded interim PK analyses will be performed for the dose escalation decisions, to select the intermediate dose for the food effect cohort, and to reconsider the sampling time points as the study progresses.

Subjects will be housed in the Celerion clinic from at least 24 hours prior (from Day -2), until 48 hours after dosing. Subjects will return for subsequent follow up safety and PK assessments on Days 4 to 7 and will be contacted via a phone call for follow-up questioning about adverse events 7 days later (Study Day 14). One cohort will return after a washout of at least 14 days or five half-lives (whichever is longer) of their fasting dose to receive the same intermediate dose (TBD mg) under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following inclusion criteria and none of the exclusion criteria to be eligible for participation in the study, unless otherwise specified. Subjects must continue to meet all inclusion criteria to be able to participate in the Food Effect study.

1. Healthy adult male and females of non-childbearing potential, 19 to 50 years of age (inclusive) at the time of screening.
2. Body mass index (BMI) ≥ 18.5 and ≤ 32.0 (kg/m2) and a body weight of no less than 50 kg.
3. Medically healthy with no clinically significant screening results (e.g., laboratory profiles, medical histories, vital signs, electrocardiograms (ECGs), physical examination) as deemed by the Principal Investigator.
4. No use of tobacco or nicotine containing products (including smoking cessation products), for a minimum of 6 months prior to dosing.
5. Females of non-childbearing potential have undergone one of the following sterilization procedures at least 6 months prior to dosing:

   i. Hysteroscopic sterilization

   ii. Bilateral tubal ligation or bilateral salpingectomy

   iii. Hysterectomy

   iv. Bilateral oophorectomy

   v. or be postmenopausal with amenorrhea for at least 1 year prior to the first dose with serumfollicle-stimulating hormone (FSH) levels consistent with postmenopausal status at screening.
6. Non-vasectomized males (or males vasectomized less than 120 days prior to study start), must agree to the following during study participation and for 90 days following the last administration of study drug:

   1. use a condom with spermicide while engaging in sexual activity or be sexually abstinent
   2. not donate sperm during this time.

   In the event the sexual partner is surgically sterile, use of a condom with spermicide is not necessary. None of the restrictions listed above are required for vasectomized males whose procedure was performed more than 120 days prior to study start.
7. Willing to answer inclusion and exclusion criteria questionnaire at check-in.
8. Subject understands study procedures and provides written informed consent for the trial.
9. Be able to comply with the protocol and the assessments therein.

Exclusion Criteria:

Subjects will be excluded from the study if there is evidence of any of the following criteria at screening or check-in, as appropriate. Subjects must continue to meet none of the Exclusion Criteria in order to participate in the Food Effect study.

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
2. History of any illness that, in the opinion of the Principal Investigator, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
3. Surgery within the past 90 days prior to dosing as determined by the Principal Investigator to be clinically relevant.
4. History or presence of alcoholism or drug abuse within the past 2 years.
5. Hypersensitive or idiosyncratic reactions to compounds related to TBA-354 (e.g., nitroimidazoles such as metronidazole, etc.).
6. Female subjects who are pregnant or lactating.
7. Positive results for the urine drug/alcohol screen at screening or check-in.
8. Positive urine cotinine at screening.
9. Positive results at screening for Human Immunodeficiency Virus (HIV), Hepatitis B Surface Antigen (HBsAg), or Hepatitis C antibodies (HCV).
10. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
11. Heart rate is lower than 40 bpm or higher than 99 bpm at screening.
12. Any clinically significant ECG abnormality at Screening (as deemed by the Principal Investigator and the Sponsor's Medical Monitor).

    NOTE: The following can be considered not clinically significant without consulting Sponsor's Medical Monitor:

    i. Mild first degree A-V block (P-R interval <0.23 sec)

    ii. Right or left axis deviation

    iii. Incomplete right bundle branch block

    iv. Isolated left anterior fascicular block (left anterior hemiblock) in younger athletic subjects
13. QTcF interval >450 msec for males or >470 msec for females (the average value for the replicate ECG at screening and Check-In), or history of prolonged QT syndrome.
14. Family history of Long-QT Syndrome or sudden death without a preceding diagnosis of a condition that could be causative of sudden death (such as known coronary artery disease, congestive heart failure or terminal cancer).
15. History of one or any combination of, the following:

    1. Seizures or seizure disorders, (excluding febrile seizures of childhood).
    2. Brain trauma or brain surgery.
    3. Any serious disorder of the CNS or related neurological system, particularly one that may lower the seizure threshold.
16. Use of any prescription medication within 14 days prior to dosing.
17. Use of any over-the-counter (OTC) medication, including herbal products and vitamins, within the 7 days prior to dosing. Up to 2 grams per day of acetaminophen is allowed at the discretion of the Principal Investigator.
18. Use of any drugs or substances known to be significant inhibitors of CYP enzymes and/or significant inhibitors or substrates of P-gp and/or OATP within 14 days prior to the first dose of study drug.
19. Use of any drugs or substances known to be inducers of CYP enzymes and/or P-gp, including St. John's Wort, within 28 days prior to the first dose of study drug.
20. Use of any drugs or substance known to lower the seizure threshold.
21. Blood donation or significant blood loss within 56 days prior to dosing.
22. Plasma donation within 7 days prior to dosing.
23. Participation in another clinical trial within 28 days prior to dosing.
24. Prior treatment with investigational products PA-824 or OPC-67683.
25. Consumption of the following prior to dosing period:

    1. Alcohol 48 hours prior to dosing
    2. Grapefruit/Mandarin Oranges 10 days prior to dosing
    3. Caffeine/Xanthine 24 hours prior to dosing

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study will be the number and severity of treatment emergent adverse events (TEAEs) following single doses of TBA-354 and placebo. | Day 1, 2, 4, 5, 6, 7, 14

SECONDARY OUTCOMES:
Pharmacokinetics of TBA-354 in plasma following single oral doses. Cmax, AUC0-24 | Day 1 (Hour 0, 1, 2, 4, 6, 7, 8, 12, 16), Day 2 (Hour 20, 24, 30, 36, 42), Follow up (Hour 72, 96, 120, 144)
  Tmax: Time of the maximum drug concentration (obtained without interpolation). Cmax: Maximum observed drug concentration. AUC0-24: Area under concentration time curve 0 to 24 hours
Effect of food on the Pharmacokinetics parameters of TBA-354 in plasma following an intermediate single oral dose. Cmax, AUC0-24 | Day 1 (Hour 0, 1, 2, 4, 6, 7, 8, 12, 16), Day 2 (Hour 20, 24, 30, 36, 42), Follow up (Hour 72, 96, 120, 144)
  Tmax: Time of the maximum drug concentration (obtained without interpolation). Cmax: Maximum observed drug concentration. AUC0-24: Area under concentration time curve 0 to 24 hours
Number of subjects/time points with abnormal findings in safety electrocardiogram | Screening; Day 1 (Hour 0, 1, 2, 4, 6, 8, 12, 16); Day 2 Hour 20, 24, 30, 36 and 48; Follow up Hour 144
  Calculated in terms of QT corrected for heart rate according to Fridericia's corrected formula (QTcF) outliers (QTcF > 450, > 480, and > 500 msec; and change-from-baseline QTcF > 30 and > 60 msec).
Placebo-corrected safety electrocardiogram Change-from-baseline heart rate | Screening; Day 1 (Hour 0, 1, 2, 4, 6, 8, 12, 16); Day 2 Hour 20, 24, 30, 36 and 48; Follow up Hour 144
  Change-from-baseline heart rate, QT corrected for heart rate according to Fridericia's corrected formula (QTcF), PR, QRS, QT, and incidence of abnormal T-wave morphology from cardiodynamic electrocardiograms extracted from the pre-specified time points.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gartner, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Lincoln, Nebraska, United States